CLINICAL TRIAL: NCT02036424
Title: A 10 Month, Single Masked, Randomized Controlled Study to Assess Anti-VEGF Alone Versus Ozurdex Given Every 3 Months for Treatment of Persistent Diabetic Macular Edema
Brief Title: Anti-Vascular Endothelial Growth Factor (Anti-VEGF) Alone Versus Ozurdex Given Every 3 Months for Treatment of Persistent Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Raj K. Maturi, MD (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Raj K. Maturi, MD, Raj K. Maturi MD, PI, Maturi, Raj K., M.D., P.C.
Organization: Maturi, Raj K., M.D., P.C. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OA 003
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Calcium Dobesilate; Dexamethasone; Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Active Comparator): 1.25 mg intravitreal injection given monthly during a 6 month period
  Interventions: Drug: Bevacizumab
- Ozurdex (Active Comparator): Dexamethasone intravitreal implant, 0.7 mg given every 3 months over 6 month period with a maximum of 3 injections
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Ozurdex — intravitreal steroid
  Other Names: Dexamethasone Intravitreal Implant
  Arms: Ozurdex
Drug: Bevacizumab — antiVEGF
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
To determine if there is visual benefit with Ozurdex treatment every three months compared to monthly anti-VEGF alone, in subjects with persistent diabetic macular edema. The investigator hypothesizes more frequent administration of Ozurdex in patients that have persistent diabetic macular edema will result in a more rapid and sustained improvement of visual acuity and/or optical coherence topography (OCT) compared to the use of anti-VEGF alone.

DETAILED DESCRIPTION:
Statistics throughout this study referred to the number of eyes rather than the number of subjects. Subjects were allowed to have both eyes in the study provided that inclusion/exclusion criteria were met. Five subjects had both eyes in the study; 45 subjects were actually enrolled, resulting in 50 study eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Male of female age 18 years or older
2. Type 1 or Type 2 diabetes
3. Best corrected visual acuity (BCVA) score of >24 and <78 letters
4. History of at least 3 anti-VEGF intravitreal injections over the past 5 months
5. Presence of macular edema defined as central subfield thickness of >340 microns on Cirrus OCT

Exclusion Criteria:

1. Anti-VEGF intravitreal treatment in the last 4 weeks
2. Intravitreal steroid treatment in the last 8 weeks or Ozurdex in the last 4 months
3. Pan retinal photocoagulation (PRP) or focal laser in the last 4 months
4. Active iris neovascularization
5. Any ocular condition in the study eye that, in the opinion of the investigator, is severe enough to compromise the study result
6. Uncontrolled systemic disease
7. Known history of intraocular pressure (IOP) elevation in response to corticosteroid treatment, that is not controlled on 2 glaucoma medications
8. Current enrollment in an investigational drug study or participation in such a study within 30 days prior to the baseline visit
9. Female patients who are pregnant, nursing or planning a pregnancy or who are of childbearing potential and not using a reliable means of contraception
10. Any condition or reason (including inability to read early treatment diabetic retinopathy study (ETDRS) chart or language barrier) that precludes the patient's ability to comply with study requirements including completion of the study
11. Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
12. Aphakia or pseudophakia with anterior chamber intraocular lens
13. Hypersensitivity to any components of Ozurdex or Avastin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Raj K. Maturi, MD, PC
Locations (1):
- Raj K Maturi MD PC, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the PI's clinical practice from January 2014 through October 2014.
Pre-assignment Details: This trial had 50 study eyes from a total of 45 participants. 5 participants had both eyes in the study.
Period: Overall Study
Arm/Group | Bevacizumab | Ozurdex
Started | 23 (23 study eyes, not number of subjects) | 27 (27 study eyes, not number of subjects)
Completed | 23 (23 study eyes, not number of subjects) | 27 (27 study eyes, not number of subjects)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 23 and 27 reflect number of study eyes in each arm rather than number of subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Ozurdex | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 9 | 16 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9) | 65 (11) | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: study eyes]
  United States | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Visual Acuity Change
Description: Visual acuity was obtained using ETDRS method and the total number of letters correct using that method was used to calculate mean visual acuity change.
Time Frame: baseline to month 7
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Bevacizumab | Ozurdex
Number analyzed (Participants) | 23 | 22
Number analyzed (eyes) | 23 | 27
ETDRS letters | 5.6 (6.1) | 5.8 (7.6)

2. Primary Outcome: Change in Optical Coherence Tomography (OCT) Central Subfield Thickness (CST) From Baseline to Month Seven
Description: Optical coherence tomography (OCT) is an established medical imaging technique that uses light to capture micrometer-resolution, three-dimensional images. The image is presented in grid form which divides that retina into sections. The center most section (CST) is used for this outcome measurement.
Time Frame: baseline to month seven
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: study eyes
Arm/Group | Bevacizumab | Ozurdex
Number analyzed (Participants) | 23 | 22
Number analyzed (study eyes) | 23 | 27
microns | -13 (105) | -122 (120)

ADVERSE EVENTS:
Description: Data entered is based on number of study eyes rather than number of participants. Systemic serious adverse events are reported based on the number of participants (45), ophthalmic AEs are based on number of study eyes (50)
Arm/Group | Bevacizumab | Ozurdex
Serious Adverse Events (participants affected / at risk) | 7/23 | 3/22
Other Adverse Events (participants affected / at risk) | 10/23 | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=23) | Ozurdex (N=22)
vitreous hemorrhage (Eye disorders) | 2 (2) | 1 (1)
cranial nerve VI palsy (Eye disorders) | 1 (1) | 0 (0)
choroidal detachment (Eye disorders) | 0 (0) | 1 (1)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
colon cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=23) | Ozurdex (N=27)
epiretinal membrane (Eye disorders) | 0 (0) | 2 (2)
vitreous syneresis (Eye disorders) | 2 (2) | 3 (3)
posterior capsule opacification (Eye disorders) | 2 (2) | 4 (4)
vitreous hemorrhage (Eye disorders) | 5 (5) | 2 (2)
worsening of cataract (Eye disorders) | 4 (4) | 7 (7)
increased intraocular pressure (Eye disorders) | 0 (0) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes